CLINICAL TRIAL: NCT03521622
Title: Effectiveness of Counseling Interventions to Modify the Stage of Behavioral Change in Risk Behaviors (Smoking and Risky Alcohol Consumption) of Patient's Candidates for Surgery at the Hospital San Ignacio. Bogotá-Colombia
Brief Title: Effectiveness of Counseling Interventions to Modify Risk Behaviors in Patients at the Hospital San Ignacio.
Acronym: EFICO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario San Ignacio (Other)
Collaborators: Pontificia Universidad Javeriana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2018/07
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Risk Behavior
Keywords: counseling; behavioral therapy; tobacco; alcohol drinking
MeSH Terms: conditions — Risk-Taking; Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- brief counseling interventions (Experimental): For smoking patients the brief intervention is 5 As model for motivated patients and 5Rs for not motivated patients.
  For risky alcohol drinkers the brief intervention is simple advise for motivated patients and brief intervention for not motivated patients.
  Interventions: Behavioral: brief counseling
- Control group (Placebo Comparator): written informative material about healthy lifestyles
  Interventions: Behavioral: brief counseling

INTERVENTIONS:
Behavioral: brief counseling — Brief counseling for motivated smoker 5 As model Brief counseling for not motivated smokers 5 Rs model Brief counseling for motivated risky drinkers simple advice Brief counseling for not motivated risky drinkers brief alcohol intervention

SUMMARY:
Randomized clinical trial that aims to determine the effectiveness of a counseling intervention to modify the stage of behavioral change in risk behaviors (smoking and risky alcohol consumption) in patients candidates for scheduled surgery or diagnostic procedures at the Hospital Universitario de San Ignacio. Bogotá-Colombia

DETAILED DESCRIPTION:
Objective: to determine the effect in the behavioral change stage of an intervention to modify risk behaviors (smoking and risky alcohol consumption) in patients candidates for scheduled surgery or diagnostic procedures at the Hospital Universitario de San Ignacio. Design: controlled clinical trial with random assignment Population: patients candidates for scheduled surgery or diagnostic procedures in surgery rooms between 19 and 64 years attending the pre-anesthetic consultation of the Hospital Universitario de San Ignacio. Interventions: brief behavioral intervention to modify risk behaviors versus information material on healthy lifestyles. Measurements: the characteristics of the study population will be described and the intervention and control groups will be compared in their basic conditions. The level of advance in the stage of change in the intervention and control arm, the proportion of people with the presence of the risk factor, as well as the decrease in the consumption of tobacco and alcohol will be compared. Expected duration: 28 months. Financing: Hospital Universitario de San Ignacio and Pontificia Universidad Javeriana. Ethical aspects: the study is adjusted to international and national standards for research projects. Under this norm, it is classified in the category of minimum risk because it is a clinical experiment with a common intervention in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* candidates for scheduled surgery with a hospital stay of 3 days or less (including ambulatory surgeries) or who attend outpatient diagnostic procedures performed in surgery rooms.
* Current smokers (any tobacco product in the last month and more than 100 cigarretes in life) or risky alcohol drinkers (more than 4 or 5 alcohol standard drinks during the last year and AUDIT score between 8-15 points)
* patients with contact information
* Patients that want to participate

Exclusion Criteria:

* People who are being treated for smoking cessation or decreased consumption of alcohol.
* People with diseases that compromise their ability to understand information or their ability to verbal communication
* Patients with dependence or abuse of alcohol or other psychoactive substances other than tobacco
* Patients in action or maintenance stages of behavioral change against their risk factor

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 440 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
the level of progress in the stage of behavioral change | one and three months after the intervention
  Stages of change of Prochaska and DiClemente

SECONDARY OUTCOMES:
proportion of smokers and risky alcohol drinker | one and three months after the intervention
  proportion of smokers and risky alcohol drinker in each arm of the study

CONTACTS AND LOCATIONS:
Overall Officials: Luz H Alba, MD, Principal Investigator — Hospital San Ignacio
Locations (1):
- Hospital Universitario de San Ignacio, Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ingrid A, Olaya L, Cuevas V, Castillo JS, Becerra N, Delgado J, Canas A, Alba LH. Effectiveness of brief counselling in a hospital setting for smoking cessation and risky alcohol drinking reduction: randomised clinical trial protocol. Rev Colomb Psiquiatr (Engl Ed). 2022 Apr-Jun;51(2):146-152. doi: 10.1016/j.rcpeng.2020.06.003. Epub 2022 Jun 16. English, Spanish. PMID 35717385
- [Derived] Almonacid I, Olaya L, Cuevas V, Castillo JS, Becerra N, Delgado J, Canas A, Alba LH. Effectiveness of Brief Counseling in a Hospital Setting for Smoking Cessation and Risky Alcohol Drinking Reduction: Randomized Clinical Trial Protocol. Rev Colomb Psiquiatr (Engl Ed). 2020 Nov 12:S0034-7450(20)30085-8. doi: 10.1016/j.rcp.2020.06.005. Online ahead of print. English, Spanish. PMID 33735015